CLINICAL TRIAL: NCT03605485
Title: The Evaluation of a Novel Nasal Pillows Mask for the Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA246
Record Dates: First submitted 2018-07-22; First posted 2018-07-30 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trial Continuous Positive Airway Pressure (CPAP) mask (Experimental): Trial nasal pillows CPAP mask
  Interventions: Device: Nasal Pillows CPAP mask

INTERVENTIONS:
Device: Nasal Pillows CPAP mask — Investigative Nasal pillows Mask to be used for OSA therapy

SUMMARY:
This investigation is a prospective, non randomized, non blinded study. This investigation is designed to evaluate the performance, comfort and ease of use with the F&P trial nasal pillows mask amongst Obstructive Sleep Apnea (OSA) participants.

DETAILED DESCRIPTION:
Visit 1 will involve the participants consented in to the trial. Participants will be fitted with the F&P trial nasal pillows mask for use in-lab.

The participant will then return the mask and have a interview, this ensures the maximum time participants will be exposed to the trial mask in lab will be in 1 night.

The mask will be returned to the Institution at the conclusion of the trial and the participant will return to their previous mask. The Institution will recruit all participants within 1 week of the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years of age)
* Able to give consent
* Apnea hypopnea Index (AHI)≥ 5 on diagnostic night
* Prescribed PAP for OSA
* Existing nasal pillows mask user

Exclusion Criteria:

* Inability to give consent
* Patients who are in a coma or a decreased level of consciousness
* Anatomical or physiological conditions making automatic positive airway pressure (APAP) therapy inappropriate (e.g. unconsolidated facial structure)
* Commercial drivers who are investigated by New Zealand Transport Agency
* Current diagnosis of carbon dioxide (CO2) retention
* Pregnant or may think they are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Ease of use | 1 night
  Subjective Questionnaire
Acceptability | 1 night
  Subjective Questionnaire

SECONDARY OUTCOMES:
Objective Leak Data | 1 night
  Data obtained from participant's device - Objective

CONTACTS AND LOCATIONS:
Overall Officials: Bhavi Ogra, Principal Investigator — Employee
Locations (1):
- Fisher & Paykel Helathcare, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No